CLINICAL TRIAL: NCT00723970
Title: Seroquel XR for the Treatment of Peri and Postmenopausal Women With Major Depressive Disorder: Impact on Mood, Physical Symptoms, Sleep and Quality of Life
Brief Title: Quetiapine Extended Release (XR) for the Treatment of Menopausal Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: D1443C00008
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2009-07

CONDITIONS: Major Depressive Disorder; Insomnia; Hot Flashes
Keywords: Major Depressive Disorder; Insomnia; Hot Flashes; Menopause; Quetiapine
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders; Hot Flashes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Use of quetiapine, flexible dose (150-300 mg/day) for 8 weeks, following a 2-week placebo lead-in phase
  Interventions: Drug: Quetiapine Extended Release

INTERVENTIONS:
Drug: Quetiapine Extended Release — Quetiapine XR, 150-300 mg QHS, for 8 weeks
  Other Names: Quetiapine extended-release (Seroquel XR)

SUMMARY:
The study was designed to examine the efficacy and tolerability of quetiapine XR for the treatment of women who suffer from depression in the context of the menopausal transition and postmenopausal years. Besides the improvement of depressive symptoms, the investigators are interested in examining the impact of this medication on vasomotor symptoms (hot flashes, night sweats), sleep and overall quality of life.

DETAILED DESCRIPTION:
The menopause transition (or perimenopause) and the early postmenopausal years are marked by intense hormone fluctuations; hormone changes are frequently accompanied by the occurrence hot flashes, night sweats and sleep disturbance. Recent epidemiologic studies also demonstrate that perimenopause is a period of greater risk for the development of depressive symptoms.

To date, serotonergic antidepressants such as paroxetine and escitalopram have shown to be efficacious for the treatment of women with depression and menopause-related symptoms. We hypothesize that the use of quetiapine for this sub-population will alleviate symptoms of depression; we also anticipate that its use may enhance quality of life and improve vasomotor symptoms - the latter possibly due to quetiapine's effect on 5HT receptors and/or due to its sleep-promoting properties (e.g., by increasing the duration of total sleep time [TST], enhancing sleep efficiency, and decreasing the number of awakenings due to hot flashes).

ELIGIBILITY:
Inclusion Criteria:

* women 40 to 60 years
* diagnosis of MDD
* perimenopausal or postmenopausal

Exclusion Criteria:

* using HRT
* using psychotropic medications
* other DSM-IV axis I diagnoses other than MDD

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Changes in depressive scores (MADRS) from baseline (after a 2-week lead-in phase) to study end | 8 weeks

SECONDARY OUTCOMES:
Changes in Menopause-related scores, based on the Greene Climacteric Scale (GCS) and Hot Flash Related daily interference Scale (HFRDIS) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claudio N Soares, MD, PhD, Principal Investigator — St. Joseph's Healthcare Hamilton, McMaster University
Locations (1):
- Women's Health Concerns Clinic (WHCC), Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Frey BN, Haber E, Mendes GC, Steiner M, Soares CN. Effects of quetiapine extended release on sleep and quality of life in midlife women with major depressive disorder. Arch Womens Ment Health. 2013 Feb;16(1):83-5. doi: 10.1007/s00737-012-0314-y. Epub 2012 Nov 11. PMID 23143411
- [Derived] Soares CN, Frey BN, Haber E, Steiner M. A pilot, 8-week, placebo lead-in trial of quetiapine extended release for depression in midlife women: impact on mood and menopause-related symptoms. J Clin Psychopharmacol. 2010 Oct;30(5):612-5. doi: 10.1097/JCP.0b013e3181f1d0f2. PMID 20814317